CLINICAL TRIAL: NCT04293757
Title: Preprocedural Imaging by Rotational Angiography in Cryoballoon Ablation for Atrial Fibrillation
Brief Title: Rotational Angiography in Cryoballoon Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Vedran Velagic, Assistant professor, MD, PhD, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA001
Record Dates: First submitted 2020-02-24; First posted 2020-03-03 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: preprocedural imaging; Atrial Fibrillation; Rotational angiography
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rotational angio (Experimental): Patients that will undergo 3D rotational angiography before cryoballoon ablation
  Interventions: Procedure: Rotational angiography
- No rotational angio (No Intervention): Patients that will receive no preprocedural imaging before cryoballoon ablation

INTERVENTIONS:
Procedure: Rotational angiography — Preprocedural imaging before ablation
  Arms: Rotational angio

SUMMARY:
There is still unresolved question weather preprocedural imaging of left atrium and pulmonary veins is needed before the pulmonary vein isolation procedure for the treatment of atrial fibrillation. The investigators are conducting a randomized study to determine if 3D rotational angiography (as a mode of preprocedural imaging) performed before the cryoballoon ablation, facilitates the procedure and has positive impact on procedure characteristics and outcomes.

DETAILED DESCRIPTION:
Around 50% of cardiac electrophysiology (EP) centers are using some kind of imaging to define left atrium and pulmonary vein anatomy before the pulmonary vein isolation (PVI) procedure. Most commonly, CT or MR are performed few days/weeks before the procedure. Three dimensional rotational angiography is least commonly used. However it has the advantage that it can be performed in the EP room just before the ablation procedure. There is still no consensus if any kind of imaging is really needed to perform safe and effective PVI.

The investigators want to determine if 3D rotational angiography (as a mode of preprocedural imaging) has positive impact on procedure safety and efficacy. Also the investigators want to compare the immediate procedure characteristics. The investigators are conducting a randomized study with 1:1 randomization and planning to enroll around 100 participants with 1 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation
* persistent atrial fibrillation
* scheduled for cryoballoon ablation

Exclusion Criteria:

* longstanding persistent atrial fibrillation
* renal failure
* contrast allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
ablation success rates | 1 year
  comparison of freedom from atrial fibrillation after ablation procedure

SECONDARY OUTCOMES:
procedure duration | 1 year
  comparison of time required to finish the ablation procedure
radiation exposure | 1 year
  comparison of radiation exposure measured in fluoroscopy time (minutes) and X ray dosage measured in mGy and mcGy/m2.
contrast expenditure | 1 year
  comparison of contrast expenditure (milliliters of contrast used) between 2 groups
complication rates | 1 year
  comparison of complication rates between 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Vedran Velagić, MD, PhD, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- KBC Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No